CLINICAL TRIAL: NCT04544280
Title: Évaluation de l'Effet d'Injections répétées de Hautes Doses de Toxine Botulique Dans le Membre inférieur de Sujets cérébrolésés Spastiques Sur Les paramètres Fonctionnels et biomécaniques de Marche
Brief Title: Effect of Repeated Injections of Higher Doses of Botulinum Toxin on Lower Limb of Spastic Hemiplegic Patients on Gait.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-18 mai-217
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: stroke; botulinum neurotoxin; spasticity; hyper-resistance; MRI; muscle structure; gait rehabilitation
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: prospective, interventional, multi-centre, open-labeled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Drug: Xeomin Injectable Product

INTERVENTIONS:
Drug: Xeomin Injectable Product — Intramuscular injection

SUMMARY:
1. To show that repeated injections of higher doses of botulinum toxin are significantly more effective than the injection of unique, lower doses, on gait function.
2. To describe the effect of repeated injections of botulinum toxin on the muscle structure in terms of volume, fat accumulation and fibrosis, by means of MRI studies

DETAILED DESCRIPTION:
1. A prospective, interventional, multi-centre, open-labeled study will be carried out. Sixty stroke patients will be recruited (from the Rehabilitation Ward of Cliniques Universitaires Saint-Luc (UCLouvain), or Centre Hospitalier Universitaire de Mont Godinne (UCLouvain), or in the out-patients clinic), if they have an indication for focal chemical denervation (by botulinum toxin injections) to treat lower limb hyper-resistance (spasticity).

   Inclusion criteria: adults (>18 years old), hemiparesis secondary to stroke, date of stroke>3 months ago, lower limb hyper-resistance responsible of gait impairment, focal chemical denervation indication, ability to walk on a treadmill.

   Exclusion criteria: aphasia or major cognitive impairments limiting the functional evaluation, neurological or orthopedic affections interfering with the studied lower limb's function, BONT injections on the lower limb during the last 3 months, contraindication to BONT injections (underlying neuromuscular disease) and no contraindication to undergo an MRI study.

   Patients will benefit from 3 sessions of botulinum toxin (Xeomeen) injections at 3 months intervals. During the first session, 400 U of Xeomeen will be injected in the lower limb of the patient (and upper limb, if needed). During the second session, 600U of Xeomeen will be injected and during the third session, 800Units of Xeomeen will be injected (in the lower limb of the patient-and upper limb, if needed-). The injections will be based on the clinical evaluation carried out by one of the investigators, who are medical doctors, specialized in Physical and Rehabilitation Medicine and have experience with hyper-resistance treatment with botulinum toxin.

   Patients will be evaluated just before, a month later and 3 months after each injection session. Functional evaluations are based on the ICF model. Impairment will be evaluated by the clinical examination (range of motion -ROM- with a hand goniometer, MAS and Tardieu scale for spasticity, Fugl-Meyer test for motor control)20; by functional evaluations (10 meters walk test, 6 minutes walk test, timed up and down the stairs test, Timed Up and Go Test) and by a 3D-Quantified Gait Analysis. The limitations in activities of daily life will be evaluated by means of the ABILOCO questionnaire. Quality of life (QoL) will be evaluated with the French version of the Short-Form Health Survey SF-3624.
2. To describe the effect of repeated injections of botulinum toxin (Xeomeen) on the muscle structure in terms of volume, fat accumulation and fibrosis, a lower limb MRI will be performed before, 1-3 days and 1 month after the 1st Xeomeen injection, and 1 month after the 3rd BONT injection, for 4 MRI studies per patient. Twenty hemiplegic subjects will be recruited. They will participate to the complete study protocol, as described for our first objective. Inclusion and exclusion criteria will be the same as previously described.

Statistical analysis: The effects of treatment on continuous variables will be assessed by a one-way (time) repeated-measures analysis of variance (Anova). Ordinal data will be assessed by a non-parametric analysis. A Chi2 test will be used to compare the distributions of qualitative variables. Testing will be performed with a p-value <0,05.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis secondary to stroke, date of stroke>3 months ago, lower limb hyper resistance responsible of gait impairment, focal chemical denervation indication, ability to walk on a treadmill

Exclusion Criteria:

* aphasia or major cognitive impairments limiting the functional evaluation, neurological or orthopedic affections interfering with the studied lower limb's function, botulinum toxin injections on the lower limb during the last 3 months, contraindication to botulinum toxin injections (underlying neuromuscular disease) and no contraindication to undergo an MRI study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Temporo-spatial parameters of gait | 7-9 months
  Improvement of temporo-spatial parameters of gait as assessed by quantified gait analysis

SECONDARY OUTCOMES:
Segmental kinematics of gait | 7-9 months
  Improvement of segmental kinematics of gait as assessed by quantified gait analysis
Energetic parameters | 7-9 months
  Improvement of energetic parameters of gait as assessed by quantified gait analysis
Muscle structure | 7-9 months
  Modification of muscle structure (volume, presence of fatty and fibrotic tissue) after repeated botulinum toxin injections as evaluated by MRI imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan STOQUART, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques Universitaire Saint Luc, Brussels
  - Cliniques Universitaires UCL Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corriveau H, Hebert R, Raiche M, Dubois MF, Prince F. Postural stability in the elderly: empirical confirmation of a theoretical model. Arch Gerontol Geriatr. 2004 Sep-Oct;39(2):163-77. doi: 10.1016/j.archger.2004.03.001. PMID 15249153
- [Background] Hirvensalo M, Rantanen T, Heikkinen E. Mobility difficulties and physical activity as predictors of mortality and loss of independence in the community-living older population. J Am Geriatr Soc. 2000 May;48(5):493-8. doi: 10.1111/j.1532-5415.2000.tb04994.x. PMID 10811541
- [Background] Brandstater ME, de Bruin H, Gowland C, Clark BM. Hemiplegic gait: analysis of temporal variables. Arch Phys Med Rehabil. 1983 Dec;64(12):583-7. PMID 6661021
- [Background] Pinzur MS, Sherman R, DiMonte-Levine P, Trimble J. Gait changes in adult onset hemiplegia. Am J Phys Med. 1987 Oct;66(5):228-37. PMID 3324770
- [Background] Olney SJ, Griffin MP, McBride ID. Temporal, kinematic, and kinetic variables related to gait speed in subjects with hemiplegia: a regression approach. Phys Ther. 1994 Sep;74(9):872-85. doi: 10.1093/ptj/74.9.872. PMID 8066114
- [Background] Stoquart G, Detrembleur C, Lejeune TM. The reasons why stroke patients expend so much energy to walk slowly. Gait Posture. 2012 Jul;36(3):409-13. doi: 10.1016/j.gaitpost.2012.03.019. Epub 2012 May 1. PMID 22555062
- [Background] Caty GD, Detrembleur C, Bleyenheuft C, Deltombe T, Lejeune TM. Effect of simultaneous botulinum toxin injections into several muscles on impairment, activity, participation, and quality of life among stroke patients presenting with a stiff knee gait. Stroke. 2008 Oct;39(10):2803-8. doi: 10.1161/STROKEAHA.108.516153. Epub 2008 Jul 17. PMID 18635841
- [Background] Wissel J, Bensmail D, Ferreira JJ, Molteni F, Satkunam L, Moraleda S, Rekand T, McGuire J, Scheschonka A, Flatau-Baque B, Simon O, Rochford ET, Dressler D, Simpson DM; TOWER study investigators. Safety and efficacy of incobotulinumtoxinA doses up to 800 U in limb spasticity: The TOWER study. Neurology. 2017 Apr 4;88(14):1321-1328. doi: 10.1212/WNL.0000000000003789. Epub 2017 Mar 10. PMID 28283596
- [Background] Minamoto VB, Suzuki KP, Bremner SN, Lieber RL, Ward SR. Dramatic changes in muscle contractile and structural properties after 2 botulinum toxin injections. Muscle Nerve. 2015 Oct;52(4):649-57. doi: 10.1002/mus.24576. Epub 2015 Jun 30. PMID 25598004
- [Derived] Selves C, Dehem S, Lejeune T, Deltombe T, Stoquart G. Effects of 3 Cycles of Increasing Botulinum Toxin Doses on Functional Parameters of Post-stroke Spastic Gait: A Prospective Cohort Study. NeuroRehabilitation. 2025 Mar;56(2):175-185. doi: 10.1177/10538135241303343. Epub 2024 Dec 24. PMID 40135684